CLINICAL TRIAL: NCT01540110
Title: Phase 2 Study of Neoadjuvant Docetaxel and Cyclophosphamide in Locally Advanced or Node Positive Primary Breast Cancer With Companion Pharmacokinetic and Pharmacogenomic Analyses
Brief Title: Study of Neoadjuvant Docetaxel and Cyclophosphamide in Locally Advanced or Node Positive Primary Breast Cancer With Companion Pharmacokinetic and Pharmacogenomic Analyses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC0907
Record Dates: First submitted 2012-01-31; First posted 2012-02-28 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: Locally Advanced or Node Positive Primary Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel + cyclophosphamide (Experimental)
  Interventions: Drug: Neoadjuvant Docetaxel and Cyclophosphamide

INTERVENTIONS:
Drug: Neoadjuvant Docetaxel and Cyclophosphamide — 5.1.1 Docetaxel Docetaxel at a dose of 75 mg/m2 will be administered by intravenous infusion over 90 minutes (AFTER completion of cyclosphosphamide 600 mg/m2) on D1 every 21 days for 6 cycles using nonpolyvinylchloride tubing.
  Standard premedication with oral dexamethasone 8 mg bd on D-1, D1 and D2 will be administered. Alternatively, intravenous dexamethasone 8 mg before docetaxel followed by oral dexamethasone 8 mg bd on D1 and D2 can be given.
  Routine prevention of chemotherapy induced emesis will be administered (see 5.2.2)
  5.1.2 Cyclophosphamide
  Cyclophosphamide 600 mg/m2 by slow intravenous infusion over 10 minutes (BEFORE docetaxel) will be administered every 21 days for 6 cycles.
  No premedications are required except for routine prevention of chemotherapy induced emesis (see 5.2.2)

SUMMARY:
Primary

The purpose of this study is to evaluate tumour pathological complete response rate after six cycles of neoadjuvant docetaxel and cyclophosphamide in an Asian population.

Secondary

To assess:

1. Pharmacokinetics (PK) and pharmacogenomics (PG) of docetaxel cyclophosphamide in Asian patients,
2. Safety and toxicity of docetaxel cyclophosphamide in Asian patients, and
3. To determine efficacy of short course (3 days) filgrastim in primary and secondary prophylaxis against febrile neutropenia in patients receiving docetaxel and cyclophosphamide.

DETAILED DESCRIPTION:
Study Design and Duration

Simon Optimal two-stage Phase II design will be used for this trial. With a null hypothesis of p0=5% and an alternative hypothesis of p1=20%, significance level, α=5% and power, (1-β)=90%, a total of 41 patients will be required, with 21 patients to be recruited for the first stage.

Hence, 21 to 41 patients will be recruited at National Cancer Centre Singapore over 36 months

Patient Sample

Patients with newly diagnosed, histological confirmed HER-2 negative clinically node positive or locally advanced (cT3-T4, N0-3 or cTx, T0-4, N2-N3) primary breast cancer without evidence of metastatic disease.

Dosage/ Dosage Form, Route and Dose Regimen

Node Positive or Locally Advanced HER2 Negative Breast Cancer proceed to Docetaxel 75 mg/m2 + Cyclophosphamide 600 mg/m2 q21 days x 6 proceed to surgery

NOTE: cyclophosphamide is administered by intravenous infusion over 10 minutes followed by docetaxel over 90 minutes Patients will receive further chemotherapy, radiotherapy, endocrine therapy and targeted therapy as per institutional guidelines after surgery.

Patients with clinical non-response after 4 cycles of docetaxel and cyclophosphamide are most unlikely to have a pathological complete response. Hence, discontinuation of study and cross over to an anthracycline based chemotherapy is allowed at that point at the discretion of the treating oncologist. These patients will be classified as pathological non complete response.

Patients with progressive disease at any time will discontinue study treatment and receive salvage therapy.

Efficacy Measurements

Pathological response will be assessed by evaluation of resected surgical specimen after completion of protocol treatment.

Safety Measurements

Vital signs, Eastern Cooperative Oncology Group (ECOG) performance status, adverse events (AEs), serial laboratory safety tests. Proportion of patients with febrile neutropenia despite primary prophylactic G-CSF will be reviewed when 6,12 ,18, 24 and 30 patients have been accrued. Increase in number of doses of primary prophylactic G-CSF will be implemented if the lower limit of the 95% confidence interval of proportion exceeds 20%.

Data Analysis

All patients who have received at least 1 dose of study treatment will be included in the safety and efficacy analyses.

Pharmacokinetic (PK), Pharmacogenetic (PG) and Correlative Studies

Consent will be obtained for future analysis of any stored preoperative tumour biopsy specimens for possible gene expression profiles predictive of docetaxel and cyclophosphamide. Patients will undergo blood sampling for docetaxel and cyclophosphamide PK studies on cycle 1 day 1 (see page 22 for detailed timing). Whole blood will be collected at baseline for genotyping for CYP3A4, CYP3A5, CYP2B6, CYP2C19, ALDH, GST, ABCB1, SLCO1B3, PXR, CAR, HNF4α genes

ALL PATIENTS WITH SERIOUS ADVERSE EVENTS MUST BE FOLLOWED UP FOR OUTCOME.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed invasive breast cancer.
* Patients must have either locally advanced (cT3-T4, N0-3 or cTx, T0-4, N2-N3) or lymph node positive breast cancer
* Age >21 years. Because no dosing or adverse event data are currently available on the use of docetaxel in patients <21 years of age, children are excluded from this study but will be eligible for future pediatric phase 2 combination trials.
* Life expectancy of greater than 10 years.
* ECOG performance status <2 (Karnofsky >60%; see Appendix A).
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >3,000/mL
  * absolute neutrophil count >1,500/mL
  * platelets >100,000/mL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance >40 mL/min for patients if creatinine levels above institutional normal
* The effects of docetaxel on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* HER2 positive breast cancer
* Metastatic breast cancer
* Patients who have had any chemotherapy or radiotherapy prior to entering the study.
* Patients receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel, cyclophosphamide, lenograstim or filgrastim.
* History of pre-existing peripheral neuropathy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because chemotherapy in general including docetaxel and cyclophosphamide used in this study are pregnancy class D agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy, breastfeeding should be discontinued if the mother is treated with chemotherapy. These potential risks may also apply to other agents used in this study.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with chemotherapy or other agents administered during the study. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
* Patients with prior malignancies are excluded except for basal cell carcinoma of the skin and carcinoma in-situ of the cervix who have received curative treatment.
* Inclusion of Women and Minorities
* Both men and women of all races and ethnic groups are eligible for this trial.
* Protocol precautions and restrictions
* Patients who are pregnant or actively breast feeding are not eligible to participate in this study as stated in 3.2.8. Female patients of child bearing potential will be required to use reliable methods of contraception for the duration of the study and until 4 weeks after the last dose of study treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-08-11; Primary Completion 2015-10-20 (Actual); Study Completion 2015-10-20 (Actual)

PRIMARY OUTCOMES:
To evaluate tumour pathological complete response rate after 6 cycles of neoadjuvant docetaxel and cyclophosphamide in Asian population | 2 years
  To evaluate tumour pathological complete response rate after 6 cycles of neoadjuvant docetaxel and cyclophosphamide in Asian population

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Dent, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore